CLINICAL TRIAL: NCT02245984
Title: Comparison Effect of Applying Paper- Based Versus Electronic Nursing Process on Clinical Competence of Undergraduate Nursing Students' of Mashhad Nursing and Midwifery School
Brief Title: Effect of Applying Paper- Based Versus Electronic Nursing Process on Clinical Competence of Nursing Student
Acronym: NP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyedreza Mazloum, Mashhad University of Medical Sciences, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 922488; 123456 (Other: UMMashhad)
Record Dates: First submitted 2014-08-20; First posted 2014-09-22 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Competence
Keywords: clinical competence, nursing process, nursing student

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paper based nursing process (Experimental): for two weeks, students in paper based nursing group will be implemented paper nursing process for patients.
  Interventions: Other: paper based nursing process
- electronic nursing process (Experimental): for two weeks students in this group will be implemented electronic nursing process for patients.
  Interventions: Other: electronic nursing process

INTERVENTIONS:
Other: paper based nursing process — for two weeks, students in paper based nursing group will be implemented paper nursing process for patients.
  Arms: paper based nursing process
Other: electronic nursing process — for each of the groups separately-training program aimed to education the nursing process and how to do it (including the definition of the nursing process, advantages and its implementation and how to collect data using patient assessment forms Gordon) in the form of workshops a day (5 hours) will be implemented. Nursing process education in the two groups will similar but two hours of the program in each groups is devoted to practical training on how to implement. After completing the training program, students learn about the nursing process will be determined in the same way. Then for two weeks, students in Group A and Group B will be implemented paper and electronic nursing process for patients.
  Arms: electronic nursing process

SUMMARY:
Compare the clinical competence of undergraduate nursing students' of mashhad nursing and midwifery school in two groups applying nursing process (paper- based versus electronic).

DETAILED DESCRIPTION:
The sample consisted of at least 30 nursing students in each of the groups A (paper-based nursing process or PNP) and B (Electronic nursing process or ENP) based on random allocation (lottery sectors) will be divided into two groups. The level of knowledge about nursing process, clinical competency and clinical decision making will evaluate by the knowledge of nursing process, Meretoja competence modified and Lauri clinical decision making questionnaires, by the investigator. Then, for each of the groups separately-training program aimed to education the nursing process and how to do it (including the definition of the nursing process, advantages and its implementation and how to collect data using patient assessment forms Gordon) in the form of workshops a day (5 hours) will be implemented. Nursing process education in the two groups will similar but two hours of the program in each groups is devoted to practical training on how to implement. After completing the training program, students learn about the nursing process will be determined in the same way. Then for two weeks, students in Group A and Group B will be implemented paper and electronic nursing process for patients and researchers will perform under your guidance will be closely monitored. Clinical competence and clinical decision making will be assessed again at the end of the course with previous method. Satisfaction of the nursing process in each group will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study
* No Experience working independently (student work, employment, etc.) as a Nurse.
* Participate in the first day of the internship program

Exclusion Criteria:

* Failure to complete course training

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
clinical competency | 2 months
  clinical competency will be measured with modified nursing competence scale(NCS)

CONTACTS AND LOCATIONS:
Overall Officials: s reza mazloum, phd, Study Director — MUMS
Locations (1):
- Ghaem hospital, Mashhad, Iran

REFERENCES:
- [Result] Meretoja R, Leino-Kilpi H, Kaira AM. Comparison of nurse competence in different hospital work environments. J Nurs Manag. 2004 Sep;12(5):329-36. doi: 10.1111/j.1365-2834.2004.00422.x. PMID 15315489
- See also: Mashhad University Medical of Sciences — http://www.mums.ac.ir